CLINICAL TRIAL: NCT01525862
Title: XprESS Maxillary Sinus Balloon Dilation Study
Brief Title: XprESS Maxillary Balloon Dilation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Entellus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2091-001
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Chronic Sinusitis; Chronic Rhinosinusitis (Diagnosis)
Keywords: Balloon sinus dilation; Balloon catheters; Sinuplasty
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Balloon sinus dilation (Experimental): Balloon dilation of the maxillary sinus using a transnasal approach.
  Interventions: Device: Balloon sinus dilation

INTERVENTIONS:
Device: Balloon sinus dilation
  Other Names: XprESS Multi-Sinus Balloon Dilation Tool

SUMMARY:
A prospective, single-arm, post approval pilot study.

DETAILED DESCRIPTION:
This study is evaluating transnasal sinus balloon dilation without tissue removal to treat the maxillary sinuses in patients with sinusitis. The study will be assessing symptomatic improvement post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age.
2. Must have uncomplicated sinusitis of the maxillary sinuses with or without anterior ethmoid disease.
3. Meet EITHER the Anthem Coverage Guideline OR BlueCross BlueShield of North Carolina Corporate Medical Policy for medically necessary functional endoscopic sinus surgery (FESS) to treat uncomplicated sinusitis.
4. Have a CT scan within 6 months prior to enrollment.
5. Be mentally and physically capable (as per physician discretion) to participate in the investigation.
6. Be willing and able to sign the study-specific informed consent prior to any study-related procedures.
7. Be willing and able to undergo balloon dilation in the clinic setting.

Exclusion Criteria:

1. Have evidence of posterior ethmoid, sphenoid or frontal sinus (excludes presence of mucous retention cysts) disease requiring endoscopic sinus surgery or balloon dilatation.
2. Have presence of features consistent with sinus fungal disease.
3. Have evidence of gross polypoid disease within any of the sinuses or within the infundibulum.
4. Require concurrent nasal surgery (eg, septoplasty, turbinate reduction, etc).
5. Have previous sinus surgery (eg, sinus surgery or balloon sinuplasty).
6. Have nasal surgery (eg, septoplasty, turbinate reduction) performed within 3 months prior to enrollment.
7. Have any anatomical anomaly (ie, severe septal deviation) preventing transnasal access to the maxillary sinus outflow tract.
8. Have a history of primary ciliary dysfunction.
9. Have hemophilia.
10. Be currently undergoing, or have undergone in the past 6 months, chemotherapy for cancer or radiation therapy in the head or neck region.
11. Have a history of cystic fibrosis.
12. Have Sampter's Triad (ie, defined as having all 3 of the following: aspirin sensitivity, asthma, and sinonasal polyposis).
13. Have known sinonasal tumors or obstructive lesions.
14. Be pregnant at the time of enrollment.
15. Be unable to stop anticoagulant medication (eg, warfarin) until the International Normalized Ratio (INR) is below 1.5.
16. Be unable to stop antiplatelet (eg, clopidogrel, aspirin, etc.) for at least 7 days prior to study procedure.
17. Be currently participating in any other drug or device clinical studies excluding postapproval or marketing registry studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Gould, MD, Principal Investigator — Synergy ENT Specialists
Locations (2):
- United States (2):
  - Entellus Medical, Plymouth, Minnesota
  - Synergy ENT Specialists, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Balloon Sinus Dilation: Balloon dilation of the maxillary sinus using a transnasal approach.
  Balloon sinus dilation
Period: Overall Study
Arm/Group | Balloon Sinus Dilation
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Balloon Sinus Dilation
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 21
Lund-Mackay score [Mean (Standard Deviation); unit: units on a scale] — The Lund-Mackay score is a method for grading chronic rhinosinusitis using CT scans. The frontal, sphenoid, maxillary, anterior ethmoid, and posterior ethmoid sinus and the ostiomeatal complex on both sides are separately assigned scores of 0 (no abnormality), 1 (partial opacification), or 2 (complete opacification).
  The ostiomeatal complex is assigned a score of either 0 (not obstructed) or 2 (obstructed). The combined score can range from 0 to 24 with higher scores indicating more sinus disease.
  units on a scale | 4.7 (3.4)
Smoking status [Count of Participants; unit: Participants]
  Nonsmokers | 19
  Smokers | 2
Allergies (year-round or seasonal) [Count of Participants; unit: Participants] | 16

OUTCOME MEASURES:

1. Primary Outcome: SNOT-20 Score
Description: The 20-item Sino-Nasal Outcomes Test (SNOT-20) is a validated patient-reported outcome measure for assessing the presence and severity of symptoms of chronic rhinosinusitis. Symptoms on the SNOT-20 survey are each rated on a scale from 0 (no problem) to 5 (problem as bad as it can be) and the 20 symptom scores are averaged to provide a total score ranging from 0 to 5. The minimal clinically important difference in the SNOT-20 has been determined to be a reduction greater or equal to 0.8 in the total SNOT-20 score.
Time Frame: Baseline and 6 months post procedure
Population: All participants with baseline and 6-month follow-up SNOT-20 assessments (matched pairs).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Balloon Sinus Dilation
Number analyzed (Participants) | 21
score on a scale
  Baseline | 2.3 (0.8)
  6-Month Follow-up | 0.8 (0.6)
Statistical Analysis 1: Comparison: Balloon Sinus Dilation; Test type: Superiority; p < 0.0001, t-test, 2 sided — P values <0.05 are considered statistically significant

2. Secondary Outcome: Recovery Time
Description: Patient-reported time from procedure to ability to return to normal daily activities.
Time Frame: 1 week post procedure
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Balloon Sinus Dilation
Number analyzed (Participants) | 21
hours | 16.1 (17.8)

3. Secondary Outcome: Procedural Pain Scores
Description: Procedure pain/discomfort on a scale of 0 (no pain) to 10 (severe pain) as reported by the participant.
Time Frame: Immediately post procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Balloon Sinus Dilation
Number analyzed (Participants) | 21
score on a scale | 1.8 (1.8)

4. Secondary Outcome: Revision Rate
Description: The number of participants who require revision sinus surgery during the study duration.
Time Frame: 6 Months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Sinus Dilation
Number analyzed (Participants) | 21
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months post procedure
Arm/Group | Balloon Sinus Dilation
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Sinus Dilation (N=21)
Complication of diabetes mellitus (Endocrine disorders) | 1 (1) — Participant was hospitalized for complications related to diabetes mellitus. The event is not related to the study device or procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less